CLINICAL TRIAL: NCT03314012
Title: First-In-Human Study for Ultrasound Based Endovascular Carotid Body Ablation in Subjects With Treatment-Resistant Hypertension: A Safety and Feasibility Study
Brief Title: First-In-Human Study Evaluating a Novel Catheter Device in Subjects With Treatment-Resistant Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cibiem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1008
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Catheter-Based Carotid Body Ablation (Experimental): All subjects undergo catheter-based ablation of the carotid body using the Cibiem Transvenous Ultrasound System (CTUS).
  Interventions: Device: Catheter-Based Carotid Body Ablation

INTERVENTIONS:
Device: Catheter-Based Carotid Body Ablation — The Cibiem Transvenous Ultrasound System (CTUS) is a catheter based device delivering ultrasound energy to ablate the carotid body. The procedure is done via a percutaneous insertion of the CTUS and advancement through the femoral vein to the jugular vein in subjects with difficult to control hypertension. The procedure duration is expected to range between 60 to 90 minutes and is performed under fluoroscopic and ultrasound image guidance.

SUMMARY:
The carotid body is located at the bifurcation of the internal and external carotid arteries. It is a chemoreceptor that plays a role in the sympathetic nervous system and in the development and maintenance of hypertension. Hypertension is a major cardiovascular risk factor and is associated with coronary artery disease, stroke, chronic kidney disease, and heart failure.

The objective of this study is to assess the effectiveness and safety of a catheter-based system to ablate the carotid body and reduce blood pressure (BP) in patients with resistant hypertension and to confirm sustainability of the treatment benefits long-term as seen following surgical CB removal.

ELIGIBILITY:
Inclusion Criteria:

* Mean office SBP ≥160 mmHg and DBP ≥90 mmHg during screen-in period
* Mean daytime systolic ABPM ≥135 mmHg during screen-in period
* Adherent to a stable drug regimen of three (3) or more anti-hypertensive medications of different classes (including one (1) diuretic), with no medication changes expected for at least six (6) months post-procedure
* No change in anti-hypertensive drug prescription (dose, number of medications, or class of medication) for at least six (6) weeks prior to enrollment
* Negative pregnancy test for women of child-bearing age
* Willingness and able to comply with follow-up requirements
* Signed informed consent

Exclusion Criteria:

* Secondary causes of hypertension
* Calculated eGFR <30mL/min/1.73m2
* History of repeated episodes of hypoglycemic unawareness
* Morbid obesity, defined as Body Mass Index >40 kg/m2
* Severe obstructive sleep apnea (AHI > 35/hr.)
* Pacemaker and/or implantable defibrillators
* History of transient ischemic accident or cerebrovascular accident during six (6) months prior to screening
* History of acute heart failure, congestive heart failure (NYHA class III-IV), myocardial infarction, unstable angina, coronary bypass or coronary angioplasty during six (6) months prior to screening
* History of ipsilateral carotid endarterectomy treatment or ipsilateral carotid artery stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by incidence of major adverse events | From procedure to one month post-procedure
  Safety assessed as the combined rate of major adverse events defined as all-causes of death, hospitalization for hypertensive crisis not related to confirmed non-adherence with anti-hypertensive medications, and any device or procedure-related serious adverse event.
Mean reduction in 24-hour ambulatory systolic and diastolic blood pressure | Baseline versus six months post-procedure

SECONDARY OUTCOMES:
Composite rate of major adverse events | At 6, 12, 18, and 24 months post-procedure
  Safety assessed as the combined rate of major adverse events defined as all-causes of death and hospitalization for hypertensive crisis not related to confirmed non-adherence with anti-hypertensive medications
Mean reduction in office systolic and diastolic blood pressure, and home systolic and diastolic blood pressure | Baseline versus 3, 6, 12, 18, and 24 months
Proportion of subjects with controlled blood pressure at 6, 12, 18, and 24 months post-procedure | At 6, 12, 18, and 24 months
  Controlled blood pressure is defined as office blood pressure <140/90 mmHg, mean 24-hr ABP <130/80 mmHg, daytime ABP <135/85 mmHg, and mean nighttime ABP <120/70 mmHg
Ventricular morphometric improvements from cardiac MRI measurements | Screening versus 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, Professor, Principal Investigator — Royal Perth Hospital
Locations (7):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Na Homolce Hospital, Prague, Czechia
- Germany (3):
  - Clinic Cardiology and Angiology II, Bad Krozingen
  - Cardiovascular Center Frankfurt (CVC Frankfurt), Frankfurt
  - Klinik für Innere Medizin III, Homburg

IPD SHARING:
Plan to Share IPD: No